CLINICAL TRIAL: NCT02146560
Title: Clinical Characteristics and Functional Outcomes of Postoperative Myocardial Injury: a Prospective Cohort Study. TEAMS (Troponin Elevation After Major Surgery) Study
Brief Title: TEAMS (Troponin Elevation After Major Surgery) Study
Acronym: TEAMS
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 13-6378-A
Record Dates: First submitted 2014-05-21; First posted 2014-05-26 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2015-11

CONDITIONS: Perioperative Myocardial Infarction; Disability
Keywords: Surgery; Non-cardiac; Elective; Adult; Patients; Troponin; Myocardial; Injury; Postoperative; Recovery; Outcome
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Background to main study question: Cardiac complications are a common cause of morbidity after non-cardiac surgery. Patients with perioperative myocardial injury (both MI, and lower levels of cardiac troponin elevation) experience higher short-term and long-term mortality. They are also at substantially increased risk of additional cardiac and non-cardiac complications. It is therefore plausible that myocardial injury adversely affects quality of life. This study will compare postoperative health-related quality of life of patients who did or did not experience perioperative myocardial injury (defined by troponin-I > 0.07ng/ml) after non-cardiac surgery

Study Design: Pilot prospective cohort study (n = 300). Population: Consecutive patients undergoing non-cardiac, non-transplant surgery at UHN.

Background to secondary study questions:

1. Clinically based risk stratification tools used in non-cardiac surgery (e.g., Revised Cardiac Risk Index) are of moderate utility and assign patients only to broad risk categories. This study will examine the usefulness of pre-operative biomarkers (BNP, HbA1c, and others) in supporting cardiac risk stratification and will address the question: Is there a set of preoperative criteria that can accurately inform the decision to monitor troponin postoperatively?
2. Intra-operative physiological derangement measured with the Surgical Apgar Score correlates with morbidity and mortality 3-months postoperatively. This study will examine the relationship between the Surgical Apgar Score; continuous non-invasively monitored intraoperative metrics of hemoglobin concentration and occult hypovolemia (Pleth Variability Index) with the Masimo Radical-7 Pulse Co-Oximeter; and the primary and secondary outcomes. This aspect of the study will address the question: Can readily available intraoperative physiological data inform the decision to monitor troponin postoperatively?
3. Quality of Recovery-40 Score evaluates (in the recovery room and at 24 hours postoperatively) the patient's subjective experience of their recovery from surgery. This metric is correlated with quality of life 3-months postop. This study will evaluate correlation between Quality of Recovery-15 Score, a valid and more efficient means of measuring recovery, and the primary and secondary outcomes.
4. Approximately 2/3 of patients who have postoperative myocardial injury are asymptomatic and have no ECG changes. Diagnosis of MI requires biomarker elevation (Troponin > 0.3ng/ml) plus clinical or ECG or imaging evidence of myocardial injury. Of the latter 3 criteria, 2 are often absent. In selected patients, this study will use trans-thoracic echocardiography, CT coronary angiography, and cardiac MRI to improve diagnostic yield and define those diagnostic modalities that are most useful in the postoperative patient.

Rationale:

Postoperative myocardial injury may negatively impact health-related quality of life. Affected patients may experience higher levels of postoperative dependency. This possibility has implications for patient rehabilitation, provincial and personal healthcare costs, as well as patients' physical, emotional and mental well-being and relationships. The public health dimension of this problem could therefore be significant. In addition, an incomplete understanding exists of how individual patient cardiac risk factors, in combination with the perioperative environment, result in myocardial injury. The diagnostic investigations that are most useful in this setting have not yet been clearly defined. Patients who fail to be rescued after experiencing postoperative complications (as distinct from failure to avoid experiencing the complication in the first instance) plays a central role in postoperative mortality. Early recognition of such patients is therefore crucial. By prospectively observing a cohort of high-risk surgical patients, this study will provide insight into how these factors interact. This will allow us to better characterize the potential predictors and features of postoperative myocardial injury. We hope that our findings will aid in the identification of patient characteristics associated with increased risks of postoperative myocardial injury, thus helping to direct diagnosis, early treatment and rescue. This study will thus potentially yield important data that will positively impact future patient care and the rational use of healthcare resources.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent
* ASA 2-4
* Age > 45
* expected length of hospital stay > 48 hours

Exclusion Criteria:

* Lack of informed consent
* ASA 5
* expected length of postoperative stay < 48 hours
* unable to take beta blockers
* unable to take intravenous contrast

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective non-cardiac non-transplant surgery
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | 6 months post-operatively
  Health-related quality of life will be evaluated with World Health Organisation Disability Assessment Schedule 2.0

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 6 months postoperative
  Myocardial Infarction (Type 1 or 2) Malignant ventricular arrhythmia (including cardiac arrest) Re-vascularisation Cardiac mortality
Mortality | 6 months postoperative
  All-cause mortality
Financial cost | In-hospital
  Healthcare-associated costs of providing care for individual patients in this study

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada